CLINICAL TRIAL: NCT00075647
Title: Phase II Trial of CCI-779 in Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: CCI-779 in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02567; MDA-2003-0530; N01CM17003 (NIH); CDR0000347405 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Adenocarcinoma of the Pancreas; Recurrent Pancreatic Cancer; Stage II Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — temsirolimus; Sirolimus

ARMS (1):
- Treatment (temsirolimus) (Experimental): Patients receive CCI-779 IV over 30 minutes once weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: temsirolimus; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: temsirolimus — Given IV
  Other Names: CCI-779; cell cycle inhibitor 779; Torisel
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy, such as CCI-779, work in different ways to stop tumor cells from dividing so they stop growing or die. This phase II trial is studying how well CCI-779 works in treating patients with locally advanced or metastatic pancreatic cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the overall survival at 6 months in patients with locally advanced or metastatic pancreatic cancer treated with CCI-779.

SECONDARY OBJECTIVES:

I. Determine time to progression, progression-free survival, overall survival, and tumor response rate in patients with measurable disease treated with this drug.

II. Correlate biomarkers of response with clinical response in patients treated with this drug.

III. Determine the safety and toxicity of this drug in these patients.

OUTLINE: This is an open-label study.

Patients receive CCI-779 IV over 30 minutes once weekly. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 13 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the pancreas

  * Locally advanced or metastatic disease
* Radiographic evidence of disease
* No known brain metastases
* Performance status - ECOG 0-2
* More than 3 months
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN (5 times ULN if liver metastases are present)
* Creatinine ≤ 1.5 mg/dL
* Creatinine clearance ≥ 50 mL/min
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Fasting serum cholesterol ≤ 350 mg/dL
* Fasting triglycerides ≤ 400 mg/dL
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness
* No concurrent prophylactic hematopoietic colony-stimulating factors
* No prior chemotherapy for metastatic pancreatic cancer
* More than 2 months since prior adjuvant or neoadjuvant chemoradiotherapy for resected pancreatic cancer

  * Must have radiographic evidence of recurrent disease
* More than 2 months since prior chemoradiotherapy for locally advanced pancreatic cancer

  * Must have radiographic evidence of disease progression
* See Chemotherapy
* See Chemotherapy
* No other concurrent investigational or commercial agents or therapies for the malignancy
* No other concurrent anticancer therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-12; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 6 months
  The method of Thall and Simon will be employed.

SECONDARY OUTCOMES:
Overall response rate defined as the number of patients who achieved CR or PR divided by the number of patients treated | Up to 2 years
  95% confidence interval will be presented
Duration of response | From the time of objective response to the time of progressive disease, assessed up to 2 years
Time to progression (TTP) | From the time of the study entry to the time of relapse or progression, assessed up to 2 years
Systemic and local adverse events assessed using the established National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) | Up to 2 years
  Descriptive statistics (mean, standard deviation, median, and range) will be displayed for relevant laboratory parameters.
Levels of PTEN, AKT, and PI3K | Up to 2 years
  Expression levels will be correlated with patient survival duration using Cox proportional hazard regression analysis
Expression and phosphorylation status of p70s6k | Up to 7 days
  Descriptive statistics will be applied to report the mean, duration of the effects on p70s6k phosphorylation.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Xiong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States